CLINICAL TRIAL: NCT01532921
Title: EASE TRICUSPID Expertise-based Assessment Study on Clinical Efficacy of Contour 3D® in TRICUSPID Valve Annuloplasty
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: EASE TRICUSPID
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2017-11

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Tricuspid Valve Repair: All patients indicated for a Tricuspid Valve (TV) repair procedure concomitantly to left-sided heart surgery, and for whom the surgeon considers the implantation of a Contour 3D® Tricuspid Annuloplasty Ring most appropriate to reconstruct the diseased valve.
  Interventions: Procedure: Tricuspid valve repair; Procedure: Left-sided heart surgery; Device: Contour 3D Tricuspid Annuloplasty Ring

INTERVENTIONS:
Procedure: Tricuspid valve repair
Procedure: Left-sided heart surgery — Tricuspid valve repair was with the study device was only warranted if concomitant left-sided heart surgery was planned
Device: Contour 3D Tricuspid Annuloplasty Ring — Contour 3D Tricuspid Annuloplasty procedure was used during the tricuspid valve repair

SUMMARY:
Few clinical evidence for the Contour 3D Tricuspid Annuloplasty Ring exists; therefore, in order to position this product on the market, a post-market release study was completed. The purpose of this study was to evaluate the hemodynamic performance of the Contour 3D® Tricuspid Annuloplasty Ring following Tricuspid Valve (TV) repair in a post-market environment.

DETAILED DESCRIPTION:
The EASE TRICUSPID Clinical Trial was a prospective, non-randomized, non-interventional, post-market release study. The purpose of this study was to evaluate the hemodynamic performance of the Contour 3D® Tricuspid Annuloplasty Ring following Tricuspid Valve (TV) repair in a post-market environment. Therefore, the primary objective of the EASE Tricuspid Study was to evaluate the hemodynamic performance of the Contour 3D® Tricuspid Annuloplasty Ring (Contour 3D ring) in subjects with tricuspid regurgitation who had a clinical indication for TV repair in a post-market use. Secondary objectives included the evaluation of the effect of TV repair with the Contour 3D ring on the right ventricular function, as well as the assessment of the effect of TV repair with the Contour 3D ring on the functional status in subjects undergoing TV repair in a post-market environment. Subjects eligible for TV repair and compliant with the enrollment criteria were considered by the Investigator for inclusion in the study. To minimize bias, enrolled subjects were followed by their own physician in accordance with the center's established practice for routine follow up. Follow-up sessions were planned at the physician's discretion. To meet the intended goals, appropriate clinical data were collected at baseline (pre-surgery), during the surgical procedure, at discharge and during the follow-up period at 6 months. Experienced echo-cardiologists evaluated the echos. At the time of enrollment it was not certain if the subject would receive a Contour 3D ring, since the surgeon might have decided during surgery that another treatment was more beneficial to the subject. In this case, the subject was terminated from the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign and date the Patient Informed Consent (PIC)
* Indicated for a concomitant surgical repair of the TV
* Willing to return to the hospital, where the implantation originally occurred, for a 6 month follow-up visit

Exclusion Criteria:

* Patients with a degenerative TV condition
* Patients with primary TV regurgitation
* Previous TV repair or replacement
* Stand-alone TV repair
* Already participating in another investigational device or drug study, possibly leading to bias and jeopardizing the scientific appropriate assessment of the study endpoints
* Life expectancy of less than one year
* Pregnant or desire to be pregnant within 12 months of the study treatment
* Under 18 years or over 85 years of age
* Patients with active endocarditis
* Patients with valvular retraction with severely reduced mobility
* Patients with a heavily calcified TV

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes all patients indicated for a TV repair procedure concomitantly to left-sided heart surgery, and for whom the surgeon considers the implantation of a Contour 3D® Tricuspid Annuloplasty Ring most appropriate to reconstruct the diseased valve. Patients with primary TV are not included, since this is often characterized by pathological leaflets for which the Contour 3D® Tricuspid Annuloplasty Ring would not be beneficial.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Lange, Prof. Dr., Principal Investigator — Deutsches Herzzentrum München
Locations (7):
- France (2):
  - Hôpital de Lyon - Hôpital Louis Pradel, Lyon
  - Centre Hospitalier de Mulhouse, Mulhouse
- Germany (3):
  - Albertinen Herz- und Gefäßzentrum, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Deutsches Herzzentrum München, Munich
- Israel (2):
  - Soroka Medical Center, Be'er Sheeva
  - Shaare Zedek Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guenzinger R, Lange RS, Riess FC, Hanke T, Bischoff N, Obadia JF, Sahar G, Bitran D, Roberts H Jr, Li S, Bolling SF. Six-Month Performance of a 3-Dimensional Annuloplasty Ring for Repair of Functional Tricuspid Regurgitation. Thorac Cardiovasc Surg. 2020 Sep;68(6):478-485. doi: 10.1055/s-0038-1673665. Epub 2018 Nov 16. PMID 30452076
- See also: Sponsor Website — http://www.medtronic.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Indicated for a TV Repair Procedure: All patients indicated for a TV repair procedure concomitantly to left-sided heart surgery, and for whom the surgeon considers the implantation of a Contour 3D® Tricuspid Annuloplasty Ring most appropriate to reconstruct the diseased valve.
Period: Overall Study
Arm/Group | Indicated for a TV Repair Procedure
Started (Enrolled and consented subjects) | 85
Implantation Procedure (Subjects with study device implanted) | 76
Discharge | 75
6 Months Follow Up | 68
Completed | 69
Not Completed | 16
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 7
Not completed — Device was explanted during procedure | 1

BASELINE CHARACTERISTICS:
Population: Baseline data include all subjects who underwent the implant procedure of the study device
Arm/Group | Indicated for a TV Repair Procedure
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 40
EuroSCORE II percentage score [Mean (Standard Deviation); unit: percentage] — EuroSCORE II (European System for Cardiac Operative Risk Evaluation) is a risk model that allows the calculation of the risk of death after a heart operation. The higher the score, the higher the risk of death after surgery. The included risk factors are: age, gender, renal impairment, extracardiac arteriopathy, poor mobility, previous cardiac surgery, chronic lung disease, active endocarditis, critical preoperative state, diabetes on insulin, NYHA-class, CCS Class 4 Angina, Left ventricular function, recent myocardial infarction, pulmonary hypertension and 3 procedure-related factors.
  percentage | 8.7 (9.4)
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina. NYHA I implies no limitations. NYHA II implies slight limitation of physical activity. NYHA III implies marked limitation of physical activity and finally, NYHA IV implies patients are Unable to carry on any physical activity without discomfort.
  Participants
    NYHA Class I | 4
    NYHA Class II | 23
    NYHA Class III | 40
    NYHA Class IV | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Gradient Across the Tricuspid Valve
Description: The mean gradient across the Tricuspid Valve (TV) measured via echocardiography at discharge (up to 5 days post-implant) through 6 months post-implant
Time Frame: At Baseline, Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Implanted cohort
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Baseline; Discharge (up to 5 Days Post-implant); 6 Months Follow-Up: All enrolled patients indicated for a TV repair procedure concomitantly to left-sided heart surgery, and for which the surgeon considers the implantation of a Contour 3D® Tricuspid Annuloplasty Ring most appropriate to reconstruct the diseased valve.
Arm/Group | Baseline | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 45 | 57 | 58
mmHg | 1.3 (0.6) | 2.0 (1.0) | 1.9 (0.9)

2. Primary Outcome: Change in the Degree of Tricuspid Regurgitation From Baseline Through Discharge (up to 5 Days Post-implant) and 6 Months Post-implant
Description: Change in the degree of tricuspid regurgitation measured via echocardiography from Baseline through 6 months post-implant. The severity of tricuspid regurgitation is graded by using several qualitative and quantitative methods. The degree of regurgitation is classified as "none", "Mild", "Moderate" or "Severe".
Time Frame: Baseline to Discharge (up to 5 days post-implant) and through 6 months post-implant
Population: Implanted cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 66 | 65
Participants
  Improved 4 grades | 7 | 7
  Improved 3 grades | 8 | 10
  Improved 2 grades | 27 | 31
  Improved 1 grade | 21 | 16
  No change | 3 | 1
  Worsened 2 grades | 0 | 0
  Worsened 3 grades | 0 | 0
  Worsened 4 grades | 0 | 0

3. Primary Outcome: Change in Tricuspid Valve (TV) Leaflet Coaptation Length From Baseline Through 6 Months Post-implant
Description: Change in the degree of TV leaflet coaptation length measured via echocardiography from Baseline through 6 months post-implant
Time Frame: Baseline to Discharge (up to 5 days post-implant) and to 6 months post-implant
Population: Implanted cohort
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 39 | 49
mm | -0.6 (4.6) | 0.0 (5.1)

4. Primary Outcome: Change in the Degree of Tricuspid Valve (TV) Leaflet Tethering Height From Baseline Through 6 Months Post-implant
Description: Change in the degree of TV leaflet tethering height measured via echocardiography from Baseline through 6 months post-implant
Time Frame: Baseline to Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Implanted cohort
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 39 | 50
mm | -0.2 (5.3) | -0.5 (5.2)

5. Secondary Outcome: Change in the Right Ventricle (RV) Diastolic Area From Baseline Through 6 Months Post-implant
Time Frame: Basline to Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Implanted Cohort
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 36 | 37
mm2 | 160.5 (481.3) | 50.0 (406.4)

6. Secondary Outcome: Change in the Tricuspid Annular Diameter Measured at Diastole From Baseline Through 6 Months Post-implant
Time Frame: Baseline to Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Data were not collected
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in the Right Ventricle (RV) Fractional Area From Baseline Through 6 Months Post-implant
Time Frame: Baseline to Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Implanted cohort
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 36 | 37
percentage of change | 1.7 (13.4) | -1.0 (17.0)

8. Secondary Outcome: Change in New York Heart Association (NYHA) Classification From Baseline Through 6 Months Post-implant
Description: The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina. NYHA I implies no limitations. NYHA II implies slight limitation of physical activity. NYHA III implies marked limitation of physical activity and finally, NYHA IV implies patients are Unable to carry on any physical activity without discomfort.
Time Frame: Baseline to Discharge (up to 5 days post-implant) and 6 months post-implant
Population: Implanted cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Discharge (up to 5 Days Post-implant) | 6 Months Follow-Up
Number analyzed (Participants) | 13 | 62
Participants
  Improved 3 classes | 0 | 3
  Improved 2 classes | 2 | 15
  Improved 1 class | 6 | 28
  No change | 4 | 13
  Worsened 1 class | 1 | 3
  Worsened 2 classes | 0 | 0
  Worsened 3 classes | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months Follow-up period
Arm/Group | Adverse Events Within 6 Months of Implant Procedure
All-Cause Mortality (participants affected / at risk) | 3/76
Serious Adverse Events (participants affected / at risk) | 45/76
Other Adverse Events (participants affected / at risk) | 46/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events Within 6 Months of Implant Procedure (N=76)
Atrioventricular Block, Complete (Cardiac disorders) | 10 (10)
Pericardial Effusion (Cardiac disorders) | 4 (4)
Acute Kidney injury (Renal and urinary disorders) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Haemorrhage (Vascular disorders) | 12 (13)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Atrial Tachycardia (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 6 (6)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 (1)
Pupils Unequal (Eye disorders) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1)
Impaired Healing (General disorders) | 1 (2)
Multi-Organ Failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 1 (1)
Ejection Fraction Decreased (Investigations) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events Within 6 Months of Implant Procedure (N=76)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Transfusion (Surgical and medical procedures) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 11 (11)
Atrial Fibrillation (Cardiac disorders) | 8 (8)
Pericardial Effusion (Cardiac disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less